CLINICAL TRIAL: NCT02194517
Title: Impact of ELKa, the Toolset for Prandial Insulin Dose Calculation on Metabolic Control in Children and Adolescent With Diabetes Type 1.
Brief Title: Impact of ELKa, the Toolset for Food Exchanges Calculation on Metabolic Control in Pediatric Diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ELKA-01
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; diet control toolset; food exchanges; CHO; FP
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (B) (No Intervention): Patients performing CHO and FP exchanges calculation with standard method.
- ELKa (A) (Experimental): Patients counting CHO and FP exchanges with ELKa toolset.
  Interventions: Device: ELKa

INTERVENTIONS:
Device: ELKa — ELKa should be used for every meal preparation. After choosing the name of particular product from the list, the program will give precise information about the amount of CHO and FP exchanges in serving. No standard calculation of exchanges need to be performed.
  Other Names: Diet Control Toolset; ElkaPlus USB Scale; Elka toolset; Elka PC application
  Arms: ELKa (A)

SUMMARY:
ELKa system is an advanced toolset which helps performing calculation of carbohydrate (CHO) and fat/protein (FP) exchanges. It consists of ELKa software including database of various meals and nutrients and ELKaPlus digital kitchen scale transmitting weight of products in a real-time to a computer via universal serial bus (USB) port. After choosing the name of particular product from the list, the program gives precise information about the amount of CHO and FP exchanges in serving.

The aim of the study is to investigate the benefit of using ELKa toolset in comparison with standard method of CHO and FP counting on metabolic control in type 1 diabetic children.

DETAILED DESCRIPTION:
A randomized, controlled, parallel, open-label 26-week clinical trial will be conducted in 106 pediatric patients with type 1 diabetes mellitus (DM). Patients will be randomly assigned into two groups: the group A (n=53) using ELKa system for food exchange counting and the group B (n= 53) using standard method.

The glycated hemoglobin levels will be measured in both groups at the beginning, after 3 and 6 months of observation. The group A also will be asked about the frequency of using the toolset. We will also assess secondary endpoints (mentioned below).

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 y
* Confirmed DM type 1
* DM for > 1 year
* HbA1c ≤ 10%
* Computer meeting ELKa system minimum requirements
* Kitchen arrangement providing enough space for computer with ELKa system
* Written informed consent

Exclusion Criteria:

* DM other than type 1
* Duration of diabetes < 1 year
* Conventional insulin therapy
* Nutritional disorders
* Celiac disease recognized in less than 4 months before inclusion
* Preceding experience with software
* Expected 21 or more consecutive days pausing in system usage
* Any medical condition, which, in the opinion of the investigator, would interfere with the evaluation of the subject

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycated hemoglobin) | 6 months

SECONDARY OUTCOMES:
HbA1c (glycated hemoglobin) | 3 months
ELKa usage frequency | 3 months
  Self-reported in questionnaire
ELKa usage frequency | 6 months
  Self-reported in questionnaire
Post- prandial glycemia | 3 months
  Mean post-prandial glycemia counted after the meal consumed between 1- 6 pm during subsequently 7- 10 days
Post- prandial glycemia | 6 months
  Mean post-prandial glycemia counted after the meal consumed between 1- 6 pm during subsequently 7- 10 days
mean diurnal glucose level | 3 months
mean diurnal glucose level | 6 months
Mean daily insulin dose [Insulin/kg/24h] | 3 months
Mean daily insulin dose [Insulin/kg/24h] | 6 months
BMI- standard deviation (BMI- sds) | 3 months
BMI- standard deviation (BMI- sds) | 6 months
Hypoglycemia episodes and severe hypoglycemia events | 3 months
  Hypoglycemia defined as glycemia below 70 mg/dl and, separately, glycemia below 50 mg/dl. Self-reported.
Hypoglycemia episodes and severe hypoglycemia events | 6 months
  Hypoglycemia defined as glycemia below 70 mg/dl and, separately, glycemia below 50 mg/dl. Self-reported.
Mean Amplitude of Glycemic Excursions (MAGE) | 3 months
  Measured in subgroup of patients with continuous glucose monitoring system (CGMS)
Mean Amplitude of Glycemic Excursions (MAGE) | 6 months
  Measured in subgroup of patients with CGMS
Glucose Area Under the Curve (AUC) | 3 months
  Measured in subgroup of patients with CGMS
Glucose Area Under the Curve (AUC) | 6 months
  Measured in subgroup of patients with CGMS

OTHER OUTCOMES:
Treatment satisfaction | 6 months
  Questionnaire regarded treatment satisfaction and wish to continuation.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, Professor, Study Chair — Medical University of Warsaw; Agnieszka Kowalska, MD, Study Director — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Kowalska A, Piechowiak K, Ramotowska A, Szypowska A. Impact of ELKa, the Electronic Device for Prandial Insulin Dose Calculation, on Metabolic Control in Children and Adolescents with Type 1 Diabetes Mellitus: A Randomized Controlled Trial. J Diabetes Res. 2017;2017:1708148. doi: 10.1155/2017/1708148. Epub 2017 Jan 23. PMID 28232949